CLINICAL TRIAL: NCT05400616
Title: Phase-II Randomized Control Trial of Nasal Microbiota Transplant Therapy in Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Brief Title: Nasal Microbiota Transfer Therapy in Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government); Monash Health (Other); Queensland University of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University of Queensland
Record Dates: First submitted 2022-05-12; First posted 2022-06-01 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: microbiota; transplant; paranasal sinuses; nasal lavage
MeSH Terms: conditions — Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Eligible patient participants will be randomly assigned to intervention or control group (1:1 ratio) as per a computer-generated randomisation schedule using permuted blocks of random sizes. The block sizes will not be disclosed, to ensure concealment.
  Both groups will receive two weeks of antibiotic treatment between recruitment and allocation to a study arm. The study team will work with each patient participant to find a suitable donor. Some patient participants will prefer a donor that is known to them other patients will prefer a donor that is an unknown volunteer. Potential donors who consent to participating in this study will be screened and be classified as donor-participants in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A biostatistician, not involved in assignment or care of the trial participants, will generate the randomisation sequence with a computerised random number generator. A research assistant, not involved in any other aspect of this study, will place the assigned treatments into sealed envelopes.
  Participants (Patients and donors) will be blinded from knowing if they are in the intervention group or the control group. The nurse and doctors attending to the participants will also be blinded. A member of the study team who will prepare the Nasal Microbiota Transplant therapy will not be masked. The person doing the analysis will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): For each nostril, the donated nasal wash sample is quiesced to 15 mls with saline Nasal Microbiota Transplant therapy.
  Interventions: Procedure: Microbiome Transplant
- Control (Placebo Comparator): For each nostril, 15 mls of saline will be used as the placebo therapy.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Microbiome Transplant — A raw microbiome, is collected from a donor without any sinonasal health problems, as a nasal lavage.
  Arms: Intervention
Procedure: Placebo — Normal saline.
  Arms: Control

SUMMARY:
Chronic Rhinosinusitis (CRS) is a chronic inflammatory condition of the nasal passage and paranasal sinuses that places significant burden on affected patients and global healthcare systems.

Current treatments for CRS such as long-term antibiotics, anti-inflammatory drugs, and surgery often reduce symptoms and signs of disease temporarily, however long-term results are much less satisfactory.

Recently, the theory of a damaged microbiome (dysbiosis) as a cause or promoting factor behind CRS has gained increasing evidence from the scientific community.

A condition of the gut with microbial dysbiosis (c.difficile) has previously employed microbiota transplant treatment with great success in long-term health outcomes. Such treatments are shown to repopulate bacterial microenvironment and restore protective commensal bacterial load.

A pilot study conducted by this study team trialed a novel intervention of a Nasal Microbiota Transplant in a small group of participants. Preliminary results suggested significantly improved CRS symptoms after treatment with a healthy donor microbiota transplant, compared to the pre-transplant baseline. The addition of a randomized-control trial with inclusion of a placebo group is the next step.

In this study, investigators aim to perform a two-arm, double-blinded, phase II randomized controlled clinical trial in order to assess the efficacy of a Nasal Microbiota Transplant against a placebo in a cohort of CRS patients without Nasal Polyps (CRSsNP).

DETAILED DESCRIPTION:
Current treatments for CRS such as long-term antibiotics, anti-inflammatory drugs, and surgery often reduce symptoms and signs of disease temporarily, however long-term results are much less satisfactory.

A microbiota therapy, as an alternative treatment to antibiotics, has the potential of improving outcomes for CRS patients long-term, whilst reducing the use of antibiotics in the community.

Several attempts of studies to define the role of microbiota of the nose and paranasal sinuses in health and disease have not yet been able to achieve a universal consensus. This is in part due to the significant inter-individual microbiota variation and complexity within humans. Such challenges have also limited the use of probiotic assemblages of one or a combination of few bacterial species in treatment of CRS.

The data derived from this study will add to our understanding of the role of the microbiome in the airways and its role in interfering with respiratory pathogens and host immunity. This is likely to have implications for CRS microbiome-based therapies, and also other potentially related respiratory conditions such as asthma, and chronic obstructive pulmonary disease (COPD).

In this study, investigators will recruit patients suffering from chronic rhinosinusitis without polyps (CRSsNP) and healthy participants that do not have a history of sinonasal disease. The sinus microbiome transplants will occur over a 2 week period, with regular follow up for up to 6-months post intervention. Main outcomes include change in disease severity, symptom severity, inflammatory changes, and microbial composition across the study period. Successful results from this trial may pave the way for a novel therapeutic for CRS patients.

This study has received ethics approval from the Royal Brisbane and Women's Health Human Resource and Ethics Committee (RBWH HREC).

ELIGIBILITY:
Inclusion criteria (patient):

* Diagnosis of Chronic Rhinosinusitis as defined by the presence of 2 or more major sinonasal symptoms (nasal blockage, nasal discharge, loss of smell, and facial pain/ fullness) for a minimum of 12 weeks
* Endoscopic confirmation of middle meatus inflammation or presence of mucopurulence, and /or CT confirmation of paranasal sinus inflammation.
* Previous nasal surgery with patent ostia to the diseased ethmoids and maxillary sinuses
* Signed written informed consent

Inclusion criteria (donor):

* No history of sinonasal or lower airway disease for the last 2 years other than the common cold.
* No clinical findings of sinonasal disease at the inclusion visit.
* Accepted as a donor by the patient.
* Signed informed consent to participate in the study.

Exclusion Criteria:

Exclusion criteria (patient):

* Aged <18 or >80 years
* Allergy to amoxicillin or clavulanate potassium and Clarithromycin.
* Excessive Nasal polyposis
* Antibiotic treatment in the last 4 weeks
* Patients with a history supporting a diagnosis of immune deficiency will be tested (Immunoglobulin A (IgA), Immunoglobulin M (IgM), Immunoglobulin G (IgG) and IgG subclasses, MBL) and /or are immunocompromised due to disease and / or medication ( e.g., insulin dependent diabetes mellitis, systemic corticosteroids)
* Patients who live with someone who is severly immunocompromised.
* Patients with cystic fibrosis or ciliary dyskinesia
* Patients who have been on an active investigational therapy within 2 months of screening
* Patients who have clinically significant laboratory abnormalities
* Patients who are pregnant, breast feeding or planning to become pregnant during the study
* Patients who are not willing to use a double barrier method of contraception during the study that is:-

  1. females must use contraceptive pill or Intra-uterine device (IUD) or similar and condoms
  2. males must use condoms and spermicidal gel
* Patients currently on any medication that may affect the results in an unpredictable manner
* The patient does not agree to comply with or is unable to meet all study requirements for the duration of the study period
* Patients deemed by the investigator to be unsuitable for participation in the study
* Patients who have had Coronavirus-19 (COVID-19) within the last month.

Exclusion criteria (donor):

* Findings in the prestudy pathogen scan that makes the donor unsuitable. Prestudy pathogen scan: Prior to first donation, the donors will be tested for HIV, Human T-lymphotropic virus 1 and 2, Hepatitis B and C, Syphilis, Tuberculosis, Herpes Simplex (HSV 1 and 2), Varicella Zoster (VZV), Cytomegalovirus (CMV), Epstein-Barr virus (EBV), Methicillin-resistant Staphylococcus aureus (MRSA) and a standard panel for sinonasal pathogens (Pneumococci, H. Influenza, Beta-streptococci and M. Catarrhalis).
* Donors who have had COVID-19 within the last 2 months.
* If the donor is positive for Herpes Simplex, CMV or EBV they will be considered unsuitable as a donor for a patient negative for the same pathogen. If the donor is positive for any other pathogen they will be considered unsuitable as a donor entirely.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sino-Nasal Outcome Test (SNOT-22) - 22 Item Questionnaire | Week 1 (Day 1) to Week 20
  Change of burden of disease as measured by the SNOT-22 (22 item sinonasal outcome test) questionnaire in patients. Each item graded 0-5.
  Minimum score 0, Maximum 105 Interpretation: Higher score indicates poorer disease control.

SECONDARY OUTCOMES:
Lund-Kennedy endoscopic assessment score | Week 1 (Day 1) to Week 20
  Change of grading of disease severity using the Lund-Kennedy endoscopy score based on clinical assessment of the middle meatus. 4-item criteria, with score of 0-2 Minimum score: 0, Maximum 8 Interpretation: Higher score indicates a higher degree of disease severity based on clinical assessment.
Characterisation of nasal microbiome in study participants | Week 1 (Day 1) to Week 20
  Change in nasal microbiome associated with clinical outcomes such as decrease in presence, absence or abundance of bacterial pathogens.
Characterisation of microbiome within effective donors as compared to ineffective donors | Week 1 (Day 1) - Week 2 (Day 9)
  Analysis of microbes (bacterial strains, viruses and fungi), and human cell types within donor specimens.
Adverse events of Participating Patients | From the day participating patients give signed consent (2-4 weeks before baseline) until the day of their End of study visit (Up to 33 weeks).
  Any adverse event
Cytokine level - Interleukin 5 or (IL-5) | Week 1 (Day 1) to Week 20
  Change of lL-5 in nasal secretion/swab markers across duration of study. Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample. Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).
Cytokine level - Interleukin 13 (IL-13) | Week 1 (Day 1) to Week 20
  Change of lL-13 in nasal secretion/swab markers across duration of study. Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample.
  Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).
Cytokine level - Interleukin 2 (IL-2) | Week 1 (Day 1) to Week 20
  Change of lL-2 in nasal secretion/swab markers across duration of study. Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample.
  Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).
Cytokine level - Interleukin 6 (IL-6) | Week 1 (Day 1) to Week 20
  Change of lL-6 in nasal secretion/swab markers across duration of study.Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample.
  Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).
Cytokine level - Interleukin 10 (IL-10) | Week 1 (Day 1) to Week 20
  Change of lL-10 in nasal secretion/swab markers across duration of study.Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample.
  Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).
Cytokine level - Interferon gamma (IFN-γ) | Week 1 (Day 1) to Week 20
  Change of IFN-Y in nasal secretion/swab markers across duration of study.Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample.
  Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).
Cytokine level - Interleukin 4 (IL-4) | Week 1 (Day 1) to Week 20
  Change of IL-4 in nasal secretion/swab markers across duration of study.Each cytokine will be quantified using a highly sensitive immunoassay which will use biotinylated antibodies specific to each cytokine to bind the cytokine molecules in the sample.
  Interactions measured on a flow cytometer and compared against its relevant standard. this will result in a measure of the total concentration of the cytokine in the sample (pg/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Anders Cervin, MD,FRACS, Study Director — University of Queensland/Royal Brisbane and Women's Hospital
Locations (3):
- Australia (3):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - University of Queensland, Brisbane, Queensland
  - Monash Health, Melbourne

IPD SHARING:
Plan to Share IPD: No
There may be a possibility to share deidentified individual outcome data upon request, if the request is in accordance with the privacy statements of this study.

REFERENCES:
- [Background] Marsh RL, Aho C, Beissbarth J, Bialasiewicz S, Binks M, Cervin A, Kirkham LS, Lemon KP, Slack MPE, Smith-Vaughan HC. Panel 4: Recent advances in understanding the natural history of the otitis media microbiome and its response to environmental pressures. Int J Pediatr Otorhinolaryngol. 2020 Mar;130 Suppl 1(Suppl 1):109836. doi: 10.1016/j.ijporl.2019.109836. Epub 2019 Dec 18. PMID 31879084
- [Background] Cho DY, Hunter RC, Ramakrishnan VR. The Microbiome and Chronic Rhinosinusitis. Immunol Allergy Clin North Am. 2020 May;40(2):251-263. doi: 10.1016/j.iac.2019.12.009. Epub 2020 Jan 16. PMID 32278449
- [Background] Psaltis AJ, Wormald PJ. Therapy of Sinonasal Microbiome in CRS: A Critical Approach. Curr Allergy Asthma Rep. 2017 Sep;17(9):59. doi: 10.1007/s11882-017-0726-x. PMID 28785927
- [Background] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599
- [Background] Mahdavinia M, Keshavarzian A, Tobin MC, Landay AL, Schleimer RP. A comprehensive review of the nasal microbiome in chronic rhinosinusitis (CRS). Clin Exp Allergy. 2016 Jan;46(1):21-41. doi: 10.1111/cea.12666. PMID 26510171
- [Background] Buckland JR, Thomas S, Harries PG. Can the Sino-nasal Outcome Test (SNOT-22) be used as a reliable outcome measure for successful septal surgery? Clin Otolaryngol Allied Sci. 2003 Feb;28(1):43-7. doi: 10.1046/j.1365-2273.2003.00663.x. PMID 12580880
- [Background] Rudmik L. Economics of Chronic Rhinosinusitis. Curr Allergy Asthma Rep. 2017 Apr;17(4):20. doi: 10.1007/s11882-017-0690-5. PMID 28337570
- [Background] Wagner Mackenzie B, Waite DW, Hoggard M, Douglas RG, Taylor MW, Biswas K. Bacterial community collapse: a meta-analysis of the sinonasal microbiota in chronic rhinosinusitis. Environ Microbiol. 2017 Jan;19(1):381-392. doi: 10.1111/1462-2920.13632. Epub 2017 Jan 18. PMID 27902866
- See also: Sinonasal Microbiome Transplant as a Therapy for Chronic Rhinosinusitis Without Nasal Polyps (CRSsNP) - pilot study — https://clinicaltrials.gov/ct2/show/NCT03122795